CLINICAL TRIAL: NCT01559324
Title: Randomized Controlled Comparison of Bifrontal and Right Unilateral ECT as to Effects on Depression, Global Cognitive Function and Biomarkers.
Brief Title: Electroconvulsive Therapy (ECT) for Elderly Patients With Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: MD Tor Magne Bjølseth (Unknown); MD Torfinn Lødøen Gaarden (Unknown)
Responsible Party: Principal Investigator, Gro Strømnes Dybedal, Ph.D.Student and Clinical Neuropsychologist, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6.2009.06 2011/02/0009
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifrontal ECT (BF) (Experimental): Formula-based low dose BF ECT
  Interventions: Device: ECT
- Right unilateral ECT (RU) (Experimental): Formula-based high-dose RU ECT
  Interventions: Device: ECT

INTERVENTIONS:
Device: ECT — Bifrontal ECT, low dosage
  Arms: Bifrontal ECT (BF)
Device: ECT — Right unilateral electrode position, high dosage
  Arms: Right unilateral ECT (RU)

SUMMARY:
ECT (electroconvulsive therapy) is mostly given to patients between the age of 60 - 85 years. There is limited evidence on the efficacy and cognitive side-effects of right unilateral (RU) and bifrontal (BF) electrode positions, the placements that are considered safe for the elderly. As far as the investigators know no randomized controlled trials (RCTs) have yet been published describing this population treated with BF or RU ECT. Non-demented depressed patients will be randomized to either method (n = 2x36). Symptom intensity, global cognitive function and biomarkers will be related to 20 healthy comparators. Testing, evaluation of depression and blood-tests are done before ECT-treatment, after a series of 6-16 ECT and 3 months after terminated ECT-treatment.

DETAILED DESCRIPTION:
Patients are assessed with Mini Mental Status Examination. Postictal reorientation time is measured. There is also a weekly rating of depression depth during the series. After the 6th ECT; Mini Mental Status Examination For a subgroup of patients; extensive blood-test samples are taken on the day of the 6th ECT.

Some of the patients receive continuation-ECT once monthly after the series. In these months patients receive treatment as usual (naturalistic observation).

ELIGIBILITY:
Inclusion Criteria:

* Major depression, either unipolar or bipolar.
* Competent to give informed consent.
* Passing a thorough physical examination

Exclusion Criteria:

* Previous ECT non - response
* ECT given during last 6 months
* Ongoing substance abuse
* Rapid cycling bipolar or schizoaffective disorder
* Parkinsons disease
* Cognitive impairment (MMSE < 24/30)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Depression | 5 months
  Hamilton depression Scale 17 items (HAM-D-17), Montgomery Åsberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Cognitive function | 5 months
Blood-tests | 5 months
  Cytokines, complement factors, BDNF, S-100-beta among others

CONTACTS AND LOCATIONS:
Overall Officials: Lars Tanum, Dr.Med., Study Director — University Hospital, Akershus
Locations (1):
- Diakonhjemmet Hospital, Department of Old Age Psychiatry, Oslo, Norway

REFERENCES:
- [Background] van der Wurff FB, Stek ML, Hoogendijk WJ, Beekman AT. The efficacy and safety of ECT in depressed older adults: a literature review. Int J Geriatr Psychiatry. 2003 Oct;18(10):894-904. doi: 10.1002/gps.944. PMID 14533122
- [Background] Tielkes CE, Comijs HC, Verwijk E, Stek ML. The effects of ECT on cognitive functioning in the elderly: a review. Int J Geriatr Psychiatry. 2008 Aug;23(8):789-95. doi: 10.1002/gps.1989. PMID 18311845
- [Background] Gardner BK, O'Connor DW. A review of the cognitive effects of electroconvulsive therapy in older adults. J ECT. 2008 Mar;24(1):68-80. doi: 10.1097/YCT.0b013e318165c7b0. PMID 18379338
- [Background] Kellner CH, Tobias KG, Wiegand J. Electrode placement in electroconvulsive therapy (ECT): A review of the literature. J ECT. 2010 Sep;26(3):175-80. doi: 10.1097/YCT.0b013e3181e48154. PMID 20562639
- [Background] Kellner CH, Knapp R, Husain MM, Rasmussen K, Sampson S, Cullum M, McClintock SM, Tobias KG, Martino C, Mueller M, Bailine SH, Fink M, Petrides G. Bifrontal, bitemporal and right unilateral electrode placement in ECT: randomised trial. Br J Psychiatry. 2010 Mar;196(3):226-34. doi: 10.1192/bjp.bp.109.066183. PMID 20194546
- [Derived] Gaarden TL, Engedal K, Benth JS, Larsen M, Lorentzen B, Mollnes TE, Bjolseth TM, Castellheim A. Exploration of 27 plasma immune markers: a cross-sectional comparison of 64 old psychiatric inpatients having unipolar major depression and 18 non-depressed old persons. BMC Geriatr. 2018 Jun 25;18(1):149. doi: 10.1186/s12877-018-0836-x. PMID 29940870
- [Derived] Bjolseth TM, Engedal K, Benth JS, Dybedal GS, Gaarden TL, Tanum L. Clinical efficacy of formula-based bifrontal versus right unilateral electroconvulsive therapy (ECT) in the treatment of major depression among elderly patients: a pragmatic, randomized, assessor-blinded, controlled trial. J Affect Disord. 2015 Apr 1;175:8-17. doi: 10.1016/j.jad.2014.12.054. Epub 2014 Dec 31. PMID 25590761